CLINICAL TRIAL: NCT05428228
Title: A Randomized, Placebo Controlled, Semi-Blind, Crossover Study to Evaluate the Effects of Two Novel Hydration Beverage Formulas on Rehydration in Healthy Adults
Brief Title: Clinical Study to Evaluate the Effects of Two Novel Hydration Beverage Formulas on Rehydration in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liquid I.V. (Other)
Collaborators: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SOW6
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Dehydration; Rehydration; Exercise Performance; Exercise Recovery; Cognitive Performance
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TP1 (Experimental): Participants will be administered TP1 during one of the experimental visits.
  Interventions: Other: TP1
- TP2 (Experimental): Participants will be administered TP2 during one of the experimental visits.
  Interventions: Other: TP2
- Placebo (Placebo Comparator): Participants will be administered placebo during one of the experimental visits.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: TP1 — Participants will be administered TP1 during one of the experimental visits.
  Arms: TP1
Other: TP2 — Participants will be administered TP2 during one of the experimental visits.
  Arms: TP2
Other: Placebo — Participants will be administered placebo during one of the experimental visits.
  Arms: Placebo

SUMMARY:
The aim of the clinical trial is to evaluate the efficacy of two novel hydration products on rehydration following exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female participants who are between 18 and 49 years of age (inclusive). Are in good general health (no active or uncontrolled diseases or conditions) and can ingest the assigned amount of fluid at each visit. Have a body mass index (BMI) between 17.0 and 29.9 kg/m2 (inclusive). Exercise regularly as per physical activity guidelines for Americans [structured exercise for a minimum of 150 cumulative minutes per week (low end) to 500 cumulative minutes of exercise per week (high-end)] and willing to maintain the same level of physical activity throughout the study period. Can maintain their exercise status at the beginning of the study throughout the study period. Can achieve a peak VO2 at screening that is at least 60% of their age and gender matched normative value per American College of Sports Medicine recommendations. Have normal or acceptable to the investigator vital signs (BP and HR) at screening. Individuals with childbearing potential: Agree to have urine pregnancy test performed on each trial day. Able to agree to the requirements and restrictions of this study, willing to give voluntary consent, able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

* Female participants who are lactating, pregnant or planning to become pregnant during the study. Carry a diagnosis of diabetes. Weigh less than or equal to 80 pounds at any visits. Answer "yes" to any of the questions asked on the screening questionnaire (Appendix 10.2.1). Have a history of a diagnosis of celiac disease, chronic pancreatitis, steatorrhea, unstable thyroid disease, major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorder (i.e., HIV/AIDS), cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit). Use any dietary supplements that may impact hydration status within the 30 days prior to the baseline visit (Familiarization Trial/Visit 2). Participants must observe a 30-day washout period of no supplementation to be eligible. Consume more than two standard alcoholic drinks per day. Use of inhalables, smokables, or the like (e.g., cigarettes, vaporizers, water pipes, or cannabis) within 30 days prior to the first dose of the study product or for the duration of the study. Have a medical condition that may impact ability to exercise or ability to ingest prescribed fluid volume. Smoking tobacco products.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Relative rehydration | Through study completion, an average of 8 weeks
  To determine the effect of the test products (TPs) on relative rehydration after exercise, as compared to placebo via percent plasma volume change and plasma osmolality

SECONDARY OUTCOMES:
Hydration status via sweat loss | Through study completion, an average of 8 weeks
  To determine the effect of the TPs on hydration status, as compared to placebo via sweat loss
Participants reported outcomes | Through study completion, an average of 8 weeks
  To determine the effect of the TPs on participant reported outcomes, as compared to placebo via bloating, exertion, exhaustion, thermal sensation, feeling of refreshment, stomach upset, and thirst

OTHER OUTCOMES:
Relative effects of dehydration and rehydration | Through study completion, an average of 8 weeks
  To explore the relative effects of dehydration and rehydration from the TPs and control on cognitive function, as compared to placebo via NIH cognitive toolbox - Flanker inhibitory control and attention testing performance
Exercise performance | Through study completion, an average of 8 weeks
  To explore the effect of the TPs on exercise performance, as compared to placebo via time to exhaustion

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- The University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No